CLINICAL TRIAL: NCT00345735
Title: Intranasal Fentanyl for the Treatment of Breakthrough Pain in Cancer Patients. A Randomised, Double-blind, Placebo-controlled, Cross-over Confirmatory Trial Testing Fentanyl and Placebo in Eight Breakthrough Pain Episodes
Brief Title: Intranasal Fentanyl for the Treatment of Breakthrough Pain in Cancer Patients (FT-017-IM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FT-017-IM; 2005-002347-82
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Cancer; Pain
Keywords: Cancer pain with breakthrough pain episodes
MeSH Terms: conditions — Neoplasms; Pain | interventions — Fentanyl

INTERVENTIONS:
Drug: Fentanyl

SUMMARY:
Primary Objective:

To demonstrate the efficacy of intranasal fentanyl in the treatment of breakthrough pain (BTP) in cancer patients.

Secondary Objective:

To explore the relationship between the response to the fentanyl dose and the stable background pain opioid dose.

ELIGIBILITY:
Inclusion Criteria:

1. Has the patient given informed consent according to local requirements before any trial-related activities? Trial-related activities are any procedures that would not have been performed during the routine management of the patient.
2. Is the patient a cancer patient with breakthrough pain?
3. Is the patient aged ≥ 18 years?
4. Has the patient received, for at least the past month, either oral morphine, oxycodone, hydromorphone, or transdermal fentanyl for treatment of background pain?
5. Is the current dose of the scheduled background pain opioid of the patient equivalent to 60-500 mg oral morphine/day or to 25-200 µg/hour transdermal fentanyl?
6. Is the background pain generally stable and on average controlled to a mild level (defined as ≤ 4 on an 11-point numerical rating scale [NRS]) by the background pain opioid?
7. Is the BTP(s) in general of such severe pain intensity that the patient judges he/she needs additional analgesics (apart from background pain medication) and does it normally last for more than 15 minutes?
8. Does the patient, in general, while using a stable fixed-schedule opioid regimen have at least three BTP episodes per week but no more than four BTP episodes per day?
9. Has the patient obtained at least partial relief of BTP(s) with his/her usual immediate-release strong opioid, i.e. oral morphine, oxycodone, hydromorphone or transmucosal fentanyl?
10. Is the life expectancy of the patient at least 3 months?
11. Is the patient able to use intranasal drugs?
12. Does the patient use adequate contraceptive precautions (contraceptive pill, implant or injection, or intrauterine device) in the trial period?
13. Does the patient have a negative pregnancy test?
14. Was the background pain, during a minimum of five of the seven days, controlled to a mild level (defined as ≤ 4 on an 11-point NRS) by the background pain opioid?
15. Did the patient have at least three BTP episodes during the seven days but no more than four BTP episodes per day?
16. Was the BTP(s) of such severe pain intensity that the patient took additional analgesics (apart from the usual background pain opioid)?

Exclusion Criteria:

1. Does the patient have a recent history of substance abuse?
2. Is the patient pregnant or nursing during the trial period?
3. Does the patient have neurological or psychiatric impairment that may compromise data collection?
4. Does the patient have severe hepatic impairment? (Investigator's judgement according to local practice.)
5. Has the patient had any recent therapy, which could potentially alter pain or response to analgesics to a degree, where the need for background pain opioid will be:

   * less than 60 mg morphine or morphine equivalents/day; or
   * less than 25 µg/hour transdermal fentanyl or the number of BTP episodes will be less than three per week during the trial period?
6. Has the patient had facial radiotherapy?
7. Has the patient been treated with a monoamine oxidase (MAO) inhibitor within the last 14 days?
8. Does the patient use methadone or buprenorphine?
9. Does the patient have impaired respiratory function to an extent which may severely increase the risk of clinically relevant respiratory depression by BTP fentanyl treatment?
10. Does the patient use drugs for intranasal administration?
11. Does the patient have a nasopharyngeal probe?
12. Is the patient known to be hypersensitive to fentanyl or to other opioids or any of their excipients?
13. Does the patient have any head injury, primary brain tumour, or other pathological conditions which could significantly increase the risk of increased intracranial pressure or impaired consciousness?
14. Is the patient concomitantly participating in any other trial with an investigational drug or device apart from cancer treatment and participation in NAF trial FT-016-IM within 30 days prior to inclusion in this trial?
15. Does the patient have pathological conditions of the nasal cavity as contraindications to intranasal fentanyl?

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference at 10 minutes (PID10) after administration

SECONDARY OUTCOMES:
Sum of pain intensity differences over the 0-60 minute time interval (SPID0-60) and General Impression (GI) with 5 point verbal rating scale at 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (1):
- Nycomed, Roskilde, Denmark